CLINICAL TRIAL: NCT06762314
Title: Comparative Clinical Study to Evaluate the Efficacy and Safety of Empagliflozin or Semaglutide in Overweight/Obese Patients With Type 1 Diabetes Inadequately Controlled by Insulin Therapy
Brief Title: Efficacy and Safety of Empagliflozin or Semaglutide in Overweight/Obese Patients With Type 1 Diabetes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mostafa Bahaa (Other)
Collaborators: Meshal Saud Alotaibi, Senior Clinical Pharmacist, King Salman Speicialist Hospital-Hail, K.S.A. (Unknown); Tanta University (Other)
Responsible Party: Sponsor-Investigator, Mostafa Bahaa, Lecturer, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tanta 145
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin; semaglutide; empagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): standard treatment group (control) that will be 35 patients who will receive multiply daily injections of insulin (basal/bolus) for 3 months.
  Interventions: Drug: Insulin
- Semaglutide group (Active Comparator): will include 35 patients who in addition to insulin (basal/bolus) will receive semaglutide 0.25 mg Sc once weekly for 1 month then increase to 0.5 mg SC once weekly for 2 months.
  Interventions: Drug: Insulin; Drug: Semaglutide
- Empaglflozin group (Active Comparator): will include 35 patients who will receive empagliflozin 10 mg orally once daily in addition to insulin (basal/bolus) for 3 months.
  Interventions: Drug: Insulin; Drug: Empagliflozin

INTERVENTIONS:
Drug: Insulin — Insulin is a naturally occurring hormone your pancreas makes that's essential for allowing your body to use sugar (glucose) for energy.
Drug: Semaglutide — Semaglutide is long acting glucagon like peptide which is parenterally administered as subcutaneous injection once weekly with a half-life of about 7 days
  Arms: Semaglutide group
Drug: Empagliflozin — Empagliflozin lowers blood glucose levels by preventing glucose reabsorption in the kidneys, thereby increasing the amount of glucose excreted in the urine
  Arms: Empaglflozin group

SUMMARY:
Type 1 Diabetes (T1DM) is a disease characterised by immune mediated destruction of the insulin-producing pancreatic beta cells. Overtime, obvious insulin deficiency develops which requires insulin therapy. T1DM accounts for about 5% to 10% of diabetes cases in Europe and United States. Currently, worldwide incidence is estimated to be around 15 per 100,000 people per year. Despite the advancement that has occurred in the field diabetes therapy, patient with T1DM still suffer from managing their disease as well as continuing to face diabetes related complications. The American Diabetes Association (ADA) recommend a goal of glycated haemoglobin (HbA1c) of < 7%. However, only 21% of adults in the United States has achieved this recommended goal. Once again, a multinational, multicentre study shows that only 24.3% of participants achieved the glycaemic target of HbA1c less than 7.0 %. Unfortunately, intensifying the insulin therapy in order to reach the targeted HbA1c can result in serious adverse effects of hypoglycaemia and weight gain which is in its turn is known risk factor for cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with type 1 diabetes for more than 1 year.
* Age 18-65 years.
* BMI ≥ 27 kg/m².
* HbA1c 7.5-10 % (58-86 mmol/mol)
* Inadequately controlled despite treatment with multiple daily injections of insulin for at least 1 year.

Exclusion Criteria:

History of medullary thyroid carcinoma or multiple endocrine neoplasia type 2 (MEN 2) syndrome; family history of multiple endocrine neoplasia, type 2A (MEN 2A), medullary thyroid cancer, or familial medullary thyroid cancer.

* Insulin pump treatment.
* Any prior use of GLP-1 RAs or dipeptidyl peptidase-4 inhibitors, any medication (except insulin) that could interfere with glycemic control or affect a subject's safety.
* An estimated glomerular filtration rate ≤ 30 mL/min/1.73 m2.
* Liver disease with raised alanine aminotransferase (AST), aspartate transaminase (ALT) or alkaline phosphatase (ALP)more than three times the upper normal range.
* History of pancreatitis.
* Gastroparesis.
* Pregnancy or lactation.
* History of alcohol or drug misuse, or any medical or psychological disorder that made the patient unsuitable for study participation.
* Acute symptomatic urinary tract infection or genital infection; chronic or recurrent (≥3 annual episodes) cystitis.
* Hypoglycaemia that required hospitalization or emergency treatment in the 3 months.
* DKA that required hospitalization or emergency treatment in the past 12 months.
* Treatment with anti-obesity drugs, weight-loss surgery or aggressive diet regimen leading to unstable body weight (based on Investigator's judgement) for the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-09-20 (Estimated); Study Completion 2028-11-20 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of this trial is the change in glycated haemoglobin from baseline after 3 months of treatment. | 3 months
  The primary outcome of this trial is the change in glycated haemoglobin from baseline after 3 months of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt